CLINICAL TRIAL: NCT03099668
Title: The Multidisciplinary Team: Truly Beneficial or Just the Flavour of the Day?A Randomized Controlled Study to Study Outcomes From MDT Care in Rheumatoid Arthritis
Brief Title: Multidisciplinary Team Care in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Centre for Health Services and Policy Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2016/00848
Record Dates: First submitted 2017-03-14; First posted 2017-04-04 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2017-03

CONDITIONS: Rheumatoid Arthritis; Multidisciplinary Communication
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: 1:1 parallel gruop allocation to multidisciplinary vs routine care
Who Masked: Outcomes Assessor
Masking Description: Joint counts at 3 and 6 months will be done by a blinded investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OSAC (Experimental): Single visit to a multidisciplinary clinic (the One Stop Arthritis Clinic, OSAC), followed by routine care
  Interventions: Other: Visit to a multidisciplinary clinic
- Routine care (No Intervention): Routine care

INTERVENTIONS:
Other: Visit to a multidisciplinary clinic — Visit to a multidisciplinary clinic
  Arms: OSAC

SUMMARY:
A randomised study of multidisciplinary care (MDT) versus routine care in patients with rheumatoid arthritis (RA). Patients with RA are randomised either to a single visit to a "one Stop Arthritis Clinic' (OSAC) or to see their usual rheumatologists. Data are collected at the baseline visit, and again at subsequent clinic visits (approximately 3 and 6 months). Outcomes such as quality of life, disease activity, physical function, disease specific knowledge, coping and self efficacy are evaluated. Assessment of comorbidities and preventative care (cancer screening, vaccinations, cardiovascular risk assessment and optimisation) are also assessed between the 2 arms.

DETAILED DESCRIPTION:
Hypotheses

1. Holistic review by a multidisciplinary team leads to improved outcomes such as improved disease activity, physical function and quality of life (QOL) in patients with rheumatoid arthritis (RA).
2. These improved outcomes are likely mediated via improvements in medication adherence, coping, disease specific knowledge and improved self-efficacy.
3. A "One Stop Arthritis Clinic" (OSAC) where patients are seen by a multidisciplinary team co-located in time and space, is an effective solution to delivering multidisciplinary care.

Specific aims Primary: To determine whether a multidisciplinary review, as compared to routine review by the treating rheumatologist, leads to improved QOL as measured by the European Quality of Life-5 Dimension 3 Level (EQ-5D) index at 6 months in patients with RA with deemed stable disease activity.

Secondary:

1. To examine the effect of the multidisciplinary review, as compared to routine rheumatologist review on RA disease activity (measured using the disease activity score in 28 joints, DAS28), pain (measured using a 100mm visual analogue scale (VAS), and physical function (measured using the modified Health Assessment Questionnaire, mHAQ).
2. To examine the effect of the multidisciplinary review, as compared to routine rheumatologist review on several secondary measures including self-efficacy (as measured using the Rheumatoid Arthritis Self Efficacy, RASE), Disease Specific Knowledge (DSK) using a Patient Knowledge Questionnaire (PKC), coping, medication adherence (using the Medication Adherence Report Scale (MARS) questionnaire, pill counts and adherence proportion percentage) and Patient Acceptable Symptom State (PASS)
3. To examine the effect of the multidisciplinary review, as compared to routine rheumatologist review on patient experience

   Background and Significance Burden of disease: Rheumatoid arthritis (RA) is a chronic disease affecting approximately 0.5 -0.7% of the population; and most common in working-age adults. Inadequately treated RA is a leading cause of disability, work loss and productivity loss due to irreversible joint damage in this relatively young group of the population, in the prime of their productive work-life.

   "Treat to Target" (T2T) approach: It has been clearly shown, that a T2T approach, in which therapy is escalated at regular intervals according to a pre-determined protocol and driven by consistent measurement of disease activity, is superior to routine care in achieving remission, and T2T is now standard of care. A validated, clinically sensitive composite disease activity measure, the DAS28 is routinely used to measure disease activity, and is a good predictor of disability. DAS28 values of <2.6 are defined as remission. About 50% of patients with early RA treated at the NUH rheumatology clinic achieve remission at 6 months (unpublished data, from the Singapore Early Arthritis Cohort).

   Multidisciplinary care: The multidisciplinary team (MDT) concept is increasingly gaining popularity and traction, and has been shown to improve outcomes in complex cancer care. Several rheumatology societies and quality standards recommend that patients with RA should have access to a multidisciplinary team consisting, at the minimum, of a specialist nurse, physiotherapist (PT), occupational therapist (OT) and podiatrist. This is based on the results of several randomized controlled trials showing the benefit of occupational therapy on grip strength, and physiotherapy on physical function and cardiovascular fitness in RA.

   The multidisciplinary "One Stop Arthritis Clinic" (OSAC) at the National University Hospital (NUH), Singapore. An OSAC was set up in the specialist outpatient clinic (SOC) at the National University Hospital (NUH) in January 2016 with the aim of providing point of care access to MDT care. Prior to the OSAC, MDT care for RA patients was sporadic, if at all. Most patients were treated solely by the physician (rheumatologist), with referral to members of the MDT on an "as needed" basis, and with appointments made on a different day, at a different location. Many patients declined the appointment due to the inconvenience of a separate visit and because they often perceived it as unnecessary.

   The OSAC team currently consists of 6 members, namely a rheumatologist, specialist nurse, PT, OT, podiatrist and medical social worker. Existing RA patients on follow up in NUH may be referred, on the discretion of their rheumatologist, to the OSAC. Consenting patients are seen at the OSAC at the next review, in lieu of their routine rheumatologist review. Preliminary patient surveys have reported excellent patient experience. As previously reported, and as per our experience, early success has come from careful planning of the logistics and organization of the clinic, along with full and equal participation of all stake-holders who share the same egalitarian values, thus avoiding conflict.

   However, there have been some barriers to OSAC referral, namely:

   (i) Cost: As outpatient specialist consultation in Singapore is typically paid out of pocket, with varying amount of government subsidization, patients pay anywhere from twice to 3 times the consultation fee to attend the OSAC as compared to a routine rheumatologist review. Therefore, cost to the patient plays a major role in health care decisions.

   (ii) Poor uptake on the part of the patients: A survey among our patients revealed that they have poor general awareness of allied health services. This is possibly because Asian cultures traditionally tend to adopt a doctor-centred care delivery, especially older patients who have experienced doctor-led consultations through most of their lives.

   Gaps in knowledge:

   i. Although the individual benefits of OT and PT interventions have been clearly shown, these have been mostly limited to intensive regimens involving multiple sessions with close supervision.17-20 The recommended "annual MDT review" has never been shown in a controlled trial to improve outcomes. The recommendation for annual MDT review is based mainly on observational studies and expert opinion.

   ii. Most trials of OT and PT were performed prior to the treat to target (T2T) era. It remains to be seen, whether with current effective treatments, an MDT review can further confer an additive benefit.

   Our study aims to fill some of these gaps by randomly assigning patients to either the OSAC or to routine rheumatologist care, and comprehensively studying outcomes in both groups.

   Methods

   Study design:

   Single centre, randomised, single-blind, controlled trial.

   Recruitment:

   Patients will be recruited from the rheumatology outpatient clinic at NUH, and informed consent will be taken for patients who are agreeable to participate. Consented patients will be randomised via a random number sequence generated by the Stata® statistical software and placed in sealed envelopes.

   Study visits:

   The study visits will be at 0, 3 and 6 months, timed to coincide with routine rheumatology clinic visits. The baseline visit will be approximately 3 months after the randomisation visit. Patients randomised to the intervention arm will be seen in the OSAC once, followed by visits to the routine rheumatology clinic at month 3 and 6. Patients in the control arm will be seen at the routine rheumatology clinic on all visits (0, 3 and 6 months).

   Data collection and follow-up: Patients will be followed for 6 months from the baseline visit (approximately 9 months from randomisation). Data will be collected by self-administered questionnaires and face to face interviews administered by a trained research nurse to both the intervention and control arms and blood will be drawn for potential future research from all participants at the baseline visit. Data on demographics, disease severity (seropositivity, presence of erosions) and disease activity using the DAS28 will be collected using a standard case report form (CRF) at baseline and at 6 months. Joint counts will be performed by either ML, PC, AS or the research nurse at the baseline visit. At the 3 month and 6-month visit, joint count will be performed by an independent assessor (a second research nurse), who is blinded to the study arm. A standardisation session will be conducted to improve inter-rater reliability between the various joint count assessors prior to commencement of the study. Physical function will be assessed according to the mHAQ and HR-QOL will be measured using the EQ-5D instrument at baseline and at 6 months. Pain score, self-efficacy, coping, adherence and disease specific knowledge will be measured at baseline, 3 months and 6 months using the VAS for pain, RASE, coping, MARS and Hennel patient knowledge questionnaires (PKC) respectively and foot pain will be measured using the Manchester Foot Disability Index (MFI). In addition, data on comorbidities, exercise frequency, smoking, alcohol, traditional medication use, vaccination status and adherence to recommended cancer screening will be collected. Laboratory tests and imaging will be done as part of the routine clinical care of patients with RA and relevant data will be abstracted from the electronic medical record. Treatment changes at each visit will be recorded. Resource utilisation in the form of number of clinic visits (including separate visits to see allied healthcare professionals), laboratory tests, imaging, prescriptions and procedures will be abstracted from the hospital billing database. Utilisation of the specialist nurse helpline will be recorded. Work status and number of days off work for both the patient and the caregiver (if any) will also be collected. Data on patient experience will be abstracted from the hospital electronic patient experience survey, which will be administered to all patients at the baseline visit.

   Primary outcome measure:

   European Quality of Life-5 Dimension 3 Level (EQ-5D) index at 6 months

   Secondary outcome measures:

   i. Proportion of patients in clinical remission or low RA disease activity (measured using the disease activity score in 28 joints, DAS28) (remission = DAS28 ≤ 2.6, low disease activity = DAS28 > 2.6 & ≤ 3.2) ii. Pain (measured using a 100mm visual analogue (VAS) scale iii. Physical function (measured using the modified Health Assessment Questionnaire, mHAQ).

   iv. Self-efficacy (measured using the Rheumatoid Arthritis Self Efficacy, RASE) v. Disease Specific Knowledge (DSK) using a Patient Knowledge Questionnaire (PKC) vi. Coping vii. Medication adherence (using the MARS questionnaire and pill count to calculate medication adherence proportion percentage) viii. Patient experience (using the standard hospital electronic patient experience survey, e-PES) ix. Foot pain (using the Manchester foot disability index, MFI) x. Proportion of patients who achieve adherence to guidelines for vaccination xi. Proportion of patients who achieve adherence to guidelines for cardiovascular risk management xii. Proportion of patients who achieve adherence to guidelines for bone health optimisation xiii. Proportion of patients who achieve adherence to guidelines for cancer screening xiv. Utilisation of healthcare resources (clinic visits, laboratory, imaging, procedures, prescriptions, calls to the nurse helpline) xv. Days off work (patient) xvi. Days off work (caregiver) xvii. Hours per week in productive paid or unpaid work (patient) xviii. Hours per week in productive paid or unpaid work (caregiver)

   Sample size calculation and feasibility:

   Using baseline values from patients seen at OSAC, the mean baseline EQ-5D index (descriptive) is 0.722 with a standard deviation (SD) of 0.156. Allowing for an alpha error of 5%, and 95% power to demonstrate a minimal clinically important improvement of 0.1 in the EQ-5D index, we would need a sample size of 128 for a 1:1 randomisation (64 in each arm). After allowing for a 10% dropout rate, we plan to recruit 140 patients (70 in each arm) to this study.

   Approximately 60 patients with RA are seen weekly at NUH. The OSAC runs once a week and has a capacity of 6 patients per clinic session. If we can randomize 8 patients per week (of which half would be randomized to the intervention arm, to be seen at OSAC), we would be able to recruit an adequate number of subjects in about 18 weeks. The consultation fee for the study participants' baseline visit (OSAC or routine rheumatology review) would be paid for through the grant funding; thus providing an incentive for patients to participate, and also overcoming the cost barrier for referral to OSAC. Follow up for all patients would be completed about 9 months after the last patient is recruited; thus the study can be completed in about 14 months.

   Statistical analysis: All analysis will be done using Stata® statistical software. The mean EQ-5D index at 6 months of patients in the intervention and control groups will be compared using the Student's t-test. Logistic regression will be used to calculate the odds of achieving a minimal clinically important difference in QOL (as measured by a 0.1 increase in the EQ-5D index) between the intervention vs. the control group while controlling for confounders such as age, gender, disease duration, disease severity (seropositivity, presence of erosions at baseline), disease activity (DAS28) and mHAQ at baseline. We will further determine whether self-efficacy, coping, adherence and DSK can improve prediction of QOL when they are added to the regression model.

   Strengths and limitations This is a randomized controlled study, thus controlling for bias in terms of allocation of patients to MDT care. Disease activity outcomes are blinded; as joint counts will be performed by a blinded assessor. The case report form is designed to be comprehensive, such that all possible outcomes of importance will be collected. Though cost-effectiveness is not one of the outcomes to be studied, the data collected are adequate to do a cost -effectiveness analysis if necessary.

   The main limitation of the study is that the patients cannot be blinded to the intervention (MDT care). This is inherent to the nature of the intervention. In addition, outcome assessors cannot be blinded to several of the outcomes, as they are determined from patient reported questionnaires; thus may be biased in favour of MDT care. Radiographic outcomes in terms of joint space narrowing and erosions are not collected as part of this study, as typically changes in these need time (≥ 1 year) and are relatively insensitive to subtle interventions such as ours. However, increasingly outcomes important to the patient are thought to be the most preferred outcomes to study, and have been shown to be predictive of radiographic damage.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatoid arthritis, at least 21 years old, being seen at the rheumatology clinic at the National University Hospital, Singapore

Exclusion Criteria:

* Patients who are pregnant, are unable to give informed consent, or have previously visited the One Stop Arthritis Clinic

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-11-17 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
European Quality of Life-5 Dimension 3 Level (EQ-5D) index at 6 months | 6 months
  Quality of life

SECONDARY OUTCOMES:
Proportion of patients in clinical remission or low RA disease activity (measured using the disease activity score in 28 joints, DAS28) (remission = DAS28 ≤ 2.6, low disease activity = DAS28 > 2.6 & ≤ 3.2) | 6 months
  Disease activity
Pain (measured using a 100mm visual analogue (VAS) scale | 3 months
  Pain
Physical function (measured using the modified Health Assessment Questionnaire, mHAQ). | 6 months
  Physical function (patient reported outcome)
Self-efficacy (measured using the Rheumatoid Arthritis Self Efficacy, RASE) | 3 months
  Self Efficacy
Disease Specific Knowledge (DSK) using a Patient Knowledge Questionnaire (PKC) | 3 months
  Disease specific knowledge
Coping - measured using a 100mm visual analogue scale answer to a single question "Considering your arthritis overall, how well did you cope (manage, deal, make do) with your disease during the last week ?" | 3 months
  Coping
Medication adherence (using the MARS questionnaire and pill count to calculate medication adherence proportion percentage) | 3 months
  Medication adherence
Patient Acceptable Symptom Score (PASS) | 6 months
  The PASS comprised the following question: "Think about all the ways your rheumatoid arthritis has affected you during the last week. If you were to remain for the next few months as you were during the last week, would this be acceptable or unacceptable to you?"
Patient experience (using the standard hospital electronic patient experience survey, e-PES) | 3 months
  patient experience
Foot pain (using the Manchester foot disability index, MFI) | 3 months
  Foot pain
Proportion of patients who achieve adherence to guidelines for vaccination | 6 months
  vaccination
Proportion of patients who achieve adherence to guidelines for cardiovascular risk management | 6 months
  Cardiovascular risk assessment
Proportion of patients who achieve adherence to guidelines for bone health optimisation | 6 months
  Bone health
Proportion of patients who achieve adherence to guidelines for cancer screening | 6 months
  Cancer screening
Utilisation of healthcare resources (clinic visits, laboratory, imaging, procedures, prescriptions, calls to the nurse helpline) measured as total dollar cost (from the hospital perspective) | 6 months
  Utilisation of resources
Days off work (patient) | 6 months
  Days off
Days off work (caregiver) | 6 months
  Days off for carer
Hours per week in productive paid or unpaid work (patient) | 6 months
  Working hours
Hours per week in productive paid or unpaid work (caregiver) | 6 months
  working hours (carer)

CONTACTS AND LOCATIONS:
Locations (1):
- Rheumatology outpatient clinic, National University Hospital, Singapore, Sinagpore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lahiri M, Cheung PPM, Dhanasekaran P, Wong SR, Yap A, Tan DSH, Chong SH, Tan CH, Santosa A, Phan P. Evaluation of a multidisciplinary care model to improve quality of life in rheumatoid arthritis: a randomised controlled trial. Qual Life Res. 2022 Jun;31(6):1749-1759. doi: 10.1007/s11136-021-03029-3. Epub 2021 Nov 6. PMID 34741249